CLINICAL TRIAL: NCT06445933
Title: The Correlation Between Vitamin B6 and Avoiding Depression in Pregnant and Peri-partum Women
Brief Title: Vitamin B6 and Depression in Pregnant and Peri-partum Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 202309090RIPA
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-03

CONDITIONS: Postpartum Depression; Heart Rate Variability
Keywords: Vitamins; Wearable devices
MeSH Terms: conditions — Depression, Postpartum | interventions — Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): After recruitment during 24-28 weeks of gestation, women would be given Vitamin B6 tablets (25mg/tablet, 75mg/day) until delivery. After delivery of the baby, the participants would be asked to take tablets(25mg/tablet, 50mg/day) up to six weeks postpartum.
  Interventions: Combination Product: Vitamin B6
- Placebo arm (Placebo Comparator): After recruitment during 24-28 weeks of gestation, women would be given three placebo tablets per day until delivery. After delivery of the baby, the participants would be asked to take two placebo tablets per day up to six weeks postpartum.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Vitamin B6 — The intervention is taking Vitamin B6 orally from recruitment around 24-28 gestational weeks to 6 weeks post-partum. 75mg/ day before delivery and 50mg/ day after delivery.
  Arms: Experimental arm
Combination Product: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
Perinatal depression is a highly prevalent and serious health issue during pregnancy. According to statistics, approximately one out of every ten postpartum women experiences this condition. Symptoms can manifest as mood fluctuations or emotional lows. Unfortunately, these symptoms are often overlooked by patients themselves or misinterpreted by others as normal adjustments to the new role of motherhood. Consequently, timely assistance and support are frequently lacking.

To address this, the investigators urgently need effective preventive measures for perinatal depression before it escalates. Recent research suggests that simple oral supplementation of vitamin B6 may help prevent and alleviate perinatal depression to some extent. Vitamin B6 plays several crucial roles in the body, including regulating neurotransmission and mental health. Therefore, it could contribute to maintaining emotional stability and psychological balance.

In contemporary times, numerous screening methods for perinatal depression involve questionnaires. However, these methods presuppose an awareness of the possibility of perinatal depression. Individuals who are unaware of these questionnaires may go undetected. Hence, our aim is to investigate whether cardiac electrophysiology results obtained through a wearable device could offer a more objective evaluation of the status of perinatal depression.

Our plan involves conducting a prospective study to delve deeper into the preventive and therapeutic effects of vitamin B6 on perinatal depression in pregnant women. Through systematic experiments and data analysis, the investigators aim to explore the impact of vitamin B6 dosage, duration, and timing of administration. Ultimately, the investigators hope to provide evidence-based recommendations and guidance for clinical practice. The investigators' goal is to offer new insights and methods to protect the mental health of expectant mothers, ensuring a pleasant and healthy pregnancy journey for each one.

DETAILED DESCRIPTION:
The total expected number of participants is 120, with 60 in the experimental group and 60 in the control group. Participants in the experimental group will take Vitamin B6, while those in the control group will take a placebo that looks similar. To ensure the credibility of the study and reduce bias, the investigators will adopt a randomized double-blind design. The target population is pregnant women aged 20-50 years, in their 28th-30th week of pregnancy. Vitamin B6 is an FDA-approved Class A drug in the United States, with no evidence of any side effects on the fetus. A baseline blood sample to measure Vitamin B6 concentration will be taken during the 28th-30th week of pregnancy, and another sample will be taken upon admission for delivery for follow-up. To avoid blood glucose affecting Vitamin B6 levels, both blood samples will be taken after an 8-hour fast. The experimental group will take three 25mg Vitamin B6 tablets daily (75mg/day) from the 28th-30th week until the end of pregnancy, and two 25mg Vitamin B6 tablets daily (50mg/day) for one month after delivery. The control group will take three placebo tablets daily from the 28th week until the end of pregnancy, and two placebo tablets daily for one month after delivery. The placebo tablets contain starch and resemble the shape of the Vitamin B6 tablets. During each prenatal visit from the 28th week until the end of pregnancy, doctors will remind participants to take their medication. An electronic system at NTU Hospital will also remind participants weekly to take their medication. Postpartum, study staff will remind participants every two weeks by phone to continue taking Vitamin B6 or placebo. Participants will complete a postpartum depression questionnaire at the 6-week follow-up visit. The results of the postpartum depression questionnaire will be analyzed in relation to Vitamin B6 intake. The investigators currently plan to use linear and logistic regression analysis to examine the association between depression scores and Vitamin B6 concentration. Other possible statistical methods include: Chi-square, independent t-test, Mann-Whitney U test, and Fisher's exact test. A p-value below 5% will be considered statistically significant. Data will be analyzed using SPSS 20.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 24-28 weeks of gestation
* Without a personal history of depression, bipolar disorder, schizophrenia, or other mental health conditions.

Exclusion Criteria:

* Allergic to Vitamin B6

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with GAD-2(General Anxiety Disorder-2) score≥3 and EPDS(Edinburgh Postnatal Depression Scale)≥10. | 22 weeks
  The investigators would like to see if participants taken Vitamin B6 would have lowered incidence of having GAD-2(General Anxiety Disorder-2) score≥3 or EPDS(Edinburgh Postnatal Depression Scale)≥10. The maximum score for the GAD-2 is 6, and the minimum is 0. A higher score indicates a greater likelihood of anxiety. The maximum score for the Edinburgh Postnatal Depression Scale (EPDS) is 30, and the minimum is 0. A higher score indicates a greater likelihood of postnatal depression.

CONTACTS AND LOCATIONS:
Overall Officials: HanYing Chen, Principal Investigator — Attending physician
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khodadad M, Bahadoran P, Kheirabadi GR, Sabzghabaee AM. Can Vitamin B6 Help to Prevent Postpartum Depression? A Randomized Controlled Trial. Int J Prev Med. 2021 Oct 19;12:136. doi: 10.4103/ijpvm.IJPVM_240_19. eCollection 2021. PMID 34912512